CLINICAL TRIAL: NCT03803384
Title: Effects of an Auto-Regulating Oxygen System Compared to Constant-Flow Oxygen During Walking in Hypoxemic COPD Patients - a Randomized Controlled Trial
Brief Title: Effects of an Auto-Regulating Oxygen System Compared to Constant-Flow Oxygen During Walking in Hypoxemic COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Professor Dr. med. Klaus Kenn, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: COPD FreeO2-Study
Record Dates: First submitted 2019-01-07; First posted 2019-01-14 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: COPD
Keywords: hypoxemia, exercise, oxygen, automatic oxygen-titration
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoxia; Motor Activity | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The Partcipant and Investigator is blinded to the type of oxygen supply (constant flow or auto-regulated flow).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT Order A and B (Experimental): First Endurance Shuttle walk test (A) with supplemental Oxygen therapy via auto-regulated oxygen flow rates (FreeO2) to maintain a oxygen saturation of 92% and second Endurance Shuttle walk (B) test with supplemental Oxygen therapy via constant oxygen flow rates
  Interventions: Other: Oxygen therapy
- ESWT Order B and A (Experimental): First Endurance Shuttle walk test (B) with supplemental Oxygen therapy via constant oxygen flow rates and second Endurance Shuttle walk (A) test with supplemental Oxygen therapy via auto-regulated oxygen flow rates (FreeO2) to maintain a oxygen saturation of 92%
  Interventions: Other: Oxygen therapy

INTERVENTIONS:
Other: Oxygen therapy — Oxygen supply during ESWT, once with the prescribed constant oxygen flow and once using an auto-regulated oxygen flow system setting the SpO2 target at 92%.

SUMMARY:
Oxygen therapy is a cornerstone in treating patients with severe chronic obstructive pulmonary disease. Usually, oxygen supplementation is delivered using constant-flow rates. Varying oxygenation levels may occur throughout patients´ changing activity. There is some evidence available that an auto-regulating oxygen flow system (FreeO2), which adjusts the oxygen flow automatically to prevent desoxygenation could be beneficial in comparison to a constant oxygen dose of 2 liter/min during walking. However, these possible benefits are unknown if the FreeO2 is compared to a constant oxygen dose according to the individual prescription. Therefore, the primary aim of this study is to investigate the effects of auto-regulated oxygen flow rates compared to constant oxygen flow rates as prescribed according to international guidelines on walking capacity in patients with COPD.

DETAILED DESCRIPTION:
Rationale:

Hypoxemia is frequently observed in COPD and thus can negatively impact exercise tolerance. Supplemental oxygen or long-term oxygen therapy is recommended to ensure that the patient is still able to manage his daily life. Usually, oxygen supplementation is delivered using constant flow rates during day- and nighttime or as needed. However, studies have shown, that auto-regulated oxygen flow systems (FreeO2) may enhance the patients endurance, lower the time in severe hypoxemia and increase the time spent within the SpO2 target range.

Aim of this study is to investigate the effects off an auto-regulated oxygen flow system in hypoxemic COPD patients on the patient´s endurance, the oxygen saturation, the pCO2 blood level as well as on heart rate and breathing frequency compared to the effects off the prescribed constant flow (according to the British Thoracic Society Guidelines for Home Oxygen Use in Adults) during an endurance shuttle walk test (ESWT). Additionally, patients experience, e.g. comfort and Preference of the Oxygen-delivery System will be documented.

Design:

This study is a randomized, controlled cross-over trial. Following an initial incremental shuttle walk test (ISWT) in order to determine the participants individual maximal walking capacity, the participant will perform 2 endurance shuttle walk tests (ESWT) at 85% of the maximal walking rate. In randomized order, the participants will perform one ESWT with constant flow as prescribed and one ESWT with the auto-regulated oxygen flow system.

ELIGIBILITY:
Inclusion Criteria:

* GOLD III/ IV
* Hypoxemia (PaO2<55 mmHg) under roomair conditions (rest or during exercise) or SpO2 <88% during exercise
* established Long-term oxygen therapy or given indication for a Long-term oxygen therapy
* Age: 40 to 80 years
* Participation in an inpatient pulmonary rehabilitation program (Schoen Klinik BGL, Germany)
* Written informed consent

Exclusion Criteria:

* Acute Exacerbation of COPD
* Clinical signs of any acute cardiac comorbidity
* Not able to walk

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Endurance time | Day 1 and Day 2
  Change of Walking Duration during the ESWT

SECONDARY OUTCOMES:
Change of oxygen saturation during the endurance shuttle walk test. | Day 1 and Day 2
  SpO2 measured by continuous transcutaneous recordung via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland).
Time to desaturation (SpO2 <=90%) and to severe desaturation (SpO2 <=85%) | Day 1 and Day 2
  SpO2 measured by continuous transcutaneous recordung via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland) and FreeO2 Device.
Change of capillary partial pressure of CO2 (pCO2) during endurance shuttle walk test | Day 1 and Day 2
  pCO2 measured by capillary blood gases taken before and after the ESWT.
Change of capillary partial pressure of O2 (pO2) during endurance shuttle walk test | Day 1 and Day 2
  pO2 measured by capillary blood gases taken before and after the ESWT.
Change of partial pressure of CO2 (pCO2) during endurance shuttle walk test | Day 1 and Day 2
  pCO2 measured by continuous transcutaneous recording via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland)
Change of heart rate during endurance shuttle walk test | Day 1 and Day 2
  Heart rate measured by continuous transcutaneous recordung via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland).
Change of breathing frequency during endurance shuttle walk test | Day 1 and Day 2
  Breathing frequency during the ESWT measured by ApneaLink Air™ (ResMed, ...)
Patients Preference due to oxygen delivery system | Day 1 and Day 2
  Patients will be asked to rate their experienced comfort after each ESWT

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Prof. Dr., Principal Investigator — Philipps University Marburg
Locations (1):
- Schoen Klinik Berchtesgadener Land, Schönau am Königssee, Bavaria, Germany

REFERENCES:
- [Background] Lellouche F, L'Her E, Bouchard PA, Brouillard C, Maltais F. Automatic Oxygen Titration During Walking in Subjects With COPD: A Randomized Crossover Controlled Study. Respir Care. 2016 Nov;61(11):1456-1464. doi: 10.4187/respcare.04406. Epub 2016 Oct 18. PMID 27794080
- [Derived] Schneeberger T, Jarosch I, Leitl D, Gloeckl R, Hitzl W, Dennis CJ, Geyer T, Criee CP, Koczulla AR, Kenn K. Automatic oxygen titration versus constant oxygen flow rates during walking in COPD: a randomised controlled, double-blind, crossover trial. Thorax. 2023 Apr;78(4):326-334. doi: 10.1136/thoraxjnl-2020-216509. Epub 2021 Oct 16. PMID 34656996